CLINICAL TRIAL: NCT01998932
Title: Clinical Study to Identify Biological Markers to Predict Wound Healing in Patients With Chronic Venous Ulceration of the Lower Limb
Brief Title: Predictive of Biomarkers of Healing in Chronic Venous Ulceration of the Lower Limb
Acronym: MOJITO
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 13HH0574; 15384 (Other: UK National Institute for Health Research (NIHR) Clinical Research Network Portfolio)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Varicose Ulcer
Keywords: Venous Ulcer; Leg Ulcer; Metabolomics; Ulcer Fluid
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human serum Human urine Human venous ulcer fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Venous Ulcer: Patients with a chronic venous ulcer defined as a wound of greater than four weeks in duration between the foot and the ankle with an Ankle Brachial Pressure Index greater than 0.85 and a colour venous duplex evidence of chronic venous insufficiency showing either reflux or obstruction.

SUMMARY:
Chronic venous ulceration of the lower limb poses a significant problem to patients and healthcare providers alike. 1% of the population of Western countries have either an open or healed chronic venous ulcer.

However, the pathophysiological abnormalities are not entirely clear in how raised venous pressure translates into the changes seen in the skin culminating in an open ulcer. The standard treatment of this condition in the United Kingdom is to undertaken compression bandaging of the lower limb.

In order to further their knowledge of venous ulceration, the investigators seek to determine the biological profile of venous ulcers over a maximum of twenty-eight weeks and by dividing the groups into healing and non-healing wounds, the investigators may be able to demonstrate a difference in the biological profile.

This work may provide insights into predicting who will respond to treatment and targets for treatment in the future.

DETAILED DESCRIPTION:
Forty patients with chronic venous ulceration of the lower limb who meet the inclusion criteria will be entered into the study and assessed over a twenty week period with assessments at week 0, 1, 2, 4, 8, 12 and 20. Urine, serum and ulcer fluid will be sampled.

If the ulcer has not healed, further assessments using an approved biological dressing will be undertaken at weeks 20, 21, 22, 23, 25 and 28 with further sampling of ulcer fluid, urine and serum.

Samples will undergo metabolic profiling using established metabolic profiling techniques developed at Imperial College.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18 years
* Chronic venous ulceration - Defined as wound of greater than four weeks in duration between the foot and the ankle with an Ankle Brachial Pressure Index greater than 0.85.
* Ulceration present for at least four weeks.
* Colour venous duplex evidence of chronic venous insufficiency showing either reflux or obstruction.

Exclusion Criteria:

* Acute infection in the studied lower limb within the last four weeks
* History of malignancy in the lower limb to be studied
* History of connective tissue disease
* Patients on medications that can cause immunosuppression - Corticosteroids, chemotherapy or radiotherapy for cancer and recombinant immunological medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic venous ulceration in London and Cambridge
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Imperial College Healthcare NHS Trust - Charing Cross Hospital, London

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic Venous Ulcer
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Venous Ulcer
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 22
Age, Continuous [Median (Full Range); unit: years] | 71 [37 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 28

OUTCOME MEASURES:

1. Primary Outcome: Identification of Biomarkers Predictive of Ulcer Healing.
Description: The primary outcome was biomarker identification via nuclear magnetic resonance spectroscopy and mass spectrometry. Outcome measure units - number of biomarkers predictive of ulcer healing.
Time Frame: 20 weeks
Population: Data from all participants was analysed, subgrouped by participants who healed and those who did not heal
Measure: Number; unit: Number of biomarkers
Arm/Group | Chronic Venous Ulcer
Number analyzed (Participants) | 28
Number of biomarkers | 9

2. Secondary Outcome: Differential Biological Response in Non Healing Ulcers Treated With a Biological Dressing.
Description: Non healing ulcers at twenty weeks will be treated in addition to standard dressing with a biological augmented dressing approved for use in the UK. This will determine if an alternative biological profile can be obtained representing a 'healing' response.
Time Frame: 8 weeks
Population: This part of the study was not performed
Arm/Group | Chronic Venous Ulcer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Chronic Venous Ulcer
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT01998932/Prot_SAP_000.pdf